CLINICAL TRIAL: NCT04541251
Title: Neoadjuvant Camrelizumab, Nab-paclitaxel and Carboplatin in Patients With Stage IB-IIIA Non-small Cell Lung Cancer (NANE-LC): A Prospective, Single-arm, Multicenter, Phase II Study
Brief Title: Neoadjuvant Camrelizumab, Nab-paclitaxel and Carboplatin in Stage IB-IIIA NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-061-001
Record Dates: First submitted 2020-02-09; First posted 2020-09-09 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer, Non-small Cell; Artificial Intelligence
Keywords: Non-small cell lung cancer; Neoadjuvant therapy; Immune checkpoint inhibitor; Major pathological response; Artificial intelligence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Nab-paclitaxel + Carboplatin (Experimental)
  Interventions: Drug: Camrelizumab + Nab-paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Camrelizumab + Nab-paclitaxel + Carboplatin — The patients will receive three cycles (one cycle is defined as every 21 days +/- 3 days) of neoadjuvant therapy with camrelizumab 200 mg, nab-paclitaxel 260 mg/m2, and carboplatin AUC 5. This will then be followed by surgery.

SUMMARY:
This prospective, single-arm, multicenter, phase II trial enrolled 40 patients who underwent surgery after three cycles of neoadjuvant therapy with camrelizumab, nab-paclitaxel, and carboplatin. The MPR is the primary endpoint, and the pCR, the complete resection rate, the objective response rate, the disease-free survival, adverse events, and quality of life are the secondary endpoints. The exploratory endpoints will be used to establish a multiomics artificial intelligence system for neoadjuvant therapy effect prediction and decision-making assistance based on radiomics, metabolism, genetic, and clinic-pathological characteristics and to explore drug resistance mechanisms.

ELIGIBILITY:
Inclusion criteria:

* The patients have stage IB-IIIA NSCLC.
* Patient ages are ≥ 18 years old, regardless of gender.
* The patients have an ECOG ps of 0-1, with a condition suitable for surgery.
* The patients have not received any anti-tumor treatment.
* The patients have adequate blood function.
* The patients have adequate organ function.
* The patients had been using an appropriate method of contraception, and there exists a negative pregnancy test (serum or urine) for women.
* The patients will give their signed informed consent.

Exclusion criteria:

* Patients who had a prior allogeneic tissue or organ transplantation.
* Patients who have multiple cancers.
* Patients who have any severe or uncontrolled systemic diseases.
* Patients with a positive test for HIV, HBV, or HCV.
* Patients with severe infection or with an infection that required antibiotic therapy.
* Patients with a history of interstitial lung disease, active tuberculosis, or autoimmune disease.
* Patients who have participated in any other clinical trials.
* Patients who are considered ineligible by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) Rate | After surgery (approximately 10 weeks)
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Evaluation of the pathological complete response (pCR) | After surgery (approximately 10 weeks)
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
Evaluation of complete resection (R0) rate | After surgery (approximately 10 weeks)
  Proportion of patients with no residual resection margin under the microscope after tumor resection
Disease free survival (DFS) | 36 months
  From the date of surgery to any of the following events: disease progression, disease recurrence or death from any cause.
Overall survival (OS) | 36 months
  From the date of participated in study to the date of death.
Objective response rate(ORR) | approximately 9 weeks
  The proportion of patients achieved complete or patial remission(Imageological) according to RECIST 1.1 prior to definitive surgery
Adverse events (AEs) | approximately 9 weeks
  The number of participants experiencing an AE will be assessed.An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined
Serious adverse events (SAEs) | approximately 9 weeks
  The number of participants experiencing an serious AE will be assessed
Qol Quality of Life | 36 months
  Quality of life asscesed by Quality of Life Questionnare-Core 30(EORTC QLQ-C30）of The European O-rganization for Reasearch and Functional Assessment of Cancer Therapy-Lung (FACT-L)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhou H, Lin L, Qin T, Ren W, Tan Y, Yang Q, Xu H, Xie X, Chen Y, Liu S, Li X, Li Z, Hu H, Yu Y, Yao H. Neoadjuvant camrelizumab, nab-paclitaxel, and carboplatin in patients with stage IB-IIIA non-small cell lung cancer (NANE-LC): a study protocol of prospective, single-arm, multicenter, phase II study. J Thorac Dis. 2021 Nov;13(11):6468-6475. doi: 10.21037/jtd-21-1022. PMID 34992825